CLINICAL TRIAL: NCT04952480
Title: Dose-escalated Adaptive Radiotherapy of Thoracic Disease for Small Cell Lung Cancer (DARTS): A Prospective Phase II Trial Evaluating Local Control of Adaptive Dose-escalated Radiotherapy
Brief Title: Dose-escalated Adaptive Radiotherapy of Thoracic Disease for Small Cell Lung Cancer
Acronym: DARTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0015
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; (Dose-escalated) Adaptive radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose-escalated adaptive chemoradiotherapy (Experimental): Concurrent with standard of care platinum doublet based chemotherapy (cisplatin + etoposide), radiation treatment plan will be delivered in three sequential phases with two scheduled replans during the treatment along with scaled dose limits for organs-at-risk: Phase 1 dose prescription = 14 Gy in 7 fractions; Phase 2 dose prescription = 10 Gy in 5 fractions starting the day after the final (7th) fraction is delivered; Phase 3 dose prescription = either a) 70 Gy in 35 fractions, or if this cannot be safely reached without exceeding the dose limit of an organ-at-risk, b) the maximum safe prescribe-able dose tolerance specified in the protocol. Either 3D conformal radiotherapy or IMRT planning and delivery techniques will be employed, including contouring relevant thoracic organs-at-risk. All CT simulation scans will be without contrast.
  Interventions: Radiation: Dose-escalated adaptive radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Dose-escalated adaptive radiotherapy — Adaptive planning of Radiation Therapy with two re-plans of the treatment field through course of therapy with the shrinking treatment fields according to tumor response to escalate dose, as allowed by dose to organs-at-risk.
Drug: Chemotherapy — Concurrent standard of care platinum doublet based therapy

SUMMARY:
The purpose of this study is to find out what effects of using adaptive radiotherapy to deliver chest radiation has on the ability to control lung cancer and side effects.

DETAILED DESCRIPTION:
This will be an open-label, single-arm, phase II study comparing dose escalated adaptive thoracic radiotherapy to historical control of standard of care single planned radiotherapy field for entire treatment course in patients with newly diagnosed limited stage small cell lung cancer eligible for concurrent chemoradiation with platinum doublet based chemotherapy, or extensive stage small cell lung cancer patients with radiation-targetable intra-thoracic disease and none or limited extra-thoracic disease that are eligible for up-front platinum doublet chemotherapy and are fit to receive concurrent radiotherapy.

The adaptive dose-escalated radiotherapy treatment plan will be delivered in three sequential phases with two scheduled replans during the treatment along with scaled dose limits for organs-at-risk. Up to 70 Gy in 35 fractions can be delivered to the disease without overdosing organs-at-risk, and treatment will last 5 - 7 weeks. Scheduled CT simulations for the replans will be at fraction 5 and fraction 10 to account for the expected rapidly shrinking tumour volumes. Participants will be followed for 24 months to investigate local failure rate, medium progression-free survival, overall survival, acute radiation toxicity, and late radiation toxicity. Follow-up after the study will be as per standard-of-care for secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Biopsy proven, newly diagnosed, untreated SCLC
* Completed standard of care staging investigations including: CT chest/abdomen/pelvis, bone scan and/or or PET-CT scan, CT head or MRI brain, or chest X-ray
* Eligible for platinum doublet chemotherapy
* Eligible for thoracic radiotherapy, which can also include ipsilateral supraclavicular lymph node disease
* Capable of providing written, informed consent prior to participation in the study. Patient's legally authorized representative (LAR) may sign on behalf of the patient.
* Able and willing to comply with protocol rules and follow-up regimen
* Performance status of ECOG 0-2
* Pulmonary function tests showing FEV-1 >1.0L and DLCO > 50% predicted
* Radiation-targetable intrathoracic disease

Exclusion Criteria:

* No intrathoracic disease seen to target with radiation
* Thoracic disease is contiguous to extra-thoracic sites, beyond ipsilateral supraclavicular lymph nodes
* Mixed histology disease
* Active serious infection requiring therapy
* Brain metastasis that has not been symptomatically stable on dexamethasone
* 4 or more sites of extrathoracic disease, even if 2 or more of these are present in the same organ system
* Previous CNS or thoracic radiotherapy
* Previous chemotherapy
* Ineligibility for platinum doublet chemotherapy
* Life expectancy of less than 3 months
* Prior thoracic surgery
* History of another primary malignancy other than cutaneous basal cell carcinoma unless disease-free for at least 5 years
* Pregnant or breast-feeding
* In LS-SCLC, patients that are not eligible for concurrent chemoradiotherapy
* In ES-SCLC, patients that are not eligible for concurrent chemoradiotherapy under the experimental arm
* CT contrast allergy or kidney disease with irreversibly low creatinine clearance inadequate for IV contrast administration (for the purposes of high quality contrast enhanced CT chest and abdomen for follow-up imaging)
* Lack of intrathoracic disease or intrathoracic disease spread not feasible to treat with adaptive radiotherapy
* Participant in development and conduct of the research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Local failure rate | The local failure rate will be assessed at the time point of 24 months.
  The time from diagnostic biopsy to documented progression of intrathoracic disease as assessed by CT or X-ray imaging.

SECONDARY OUTCOMES:
Progression-free survival | Median time to PFS in study population. Expected to be within 24 months.
  Time from diagnostic biopsy to first documented clinical or radiographic evidence of local progression or new metastatic disease.
Overall survival | Median time to OS in study population. Expected to be within 24 months.
  Time from diagnostic biopsy to death of the patient.
Acute radiation toxicity | Expected to be within 3 months.
  Toxicity during and in the 3 months after radiotherapy as defined by CTCAE v.5 for esophagus, skin, lung, heart, and subcutaneous tissue.
Late radiation toxicity | Late toxicity will be assessed up to 24 months post-treatment.
  Toxicity seen 3 months after radiotherapy as defined by CTCAE v.5 for esophagus, skin, lung, heart, and subcutaneous tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Don, MD, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No